CLINICAL TRIAL: NCT04052295
Title: Clinical and Sonographic Evaluation of the Diaphragm After Plication in Adults With Unilateral Eventration: a Retrospective Study
Brief Title: Clinical and Sonographic Diaphragm Evaluation Post-plication
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Bary Ahmed Ibrahim, Associate professor, South Valley University
Other Study IDs: South Valley University 1576
Record Dates: First submitted 2019-07-24; First posted 2019-08-09 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Diaphragmatic Plication; Unilateral Diaphragmatic Paralysis; Diaphragm Ultrasonography
Keywords: Diaphragmatic eventration; Diaphragm; Dyspnea
MeSH Terms: conditions — Diaphragmatic Eventration; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical diaphragmatic plication — The plication was done by the same surgeon either via a 7-8 cm long lateral thoracotomy and entrance to the pleural cavity through the eighth intercostals space on the affected side or using VATS (video-assisted thoracoscopic surgery) procedure. It was performed under single lumen intubation general anaesthesia. The diaphragm with the abdominal content was pushed caudally till the normal position of the copula achieved. At this position a fold of about 5 cm is made using traction forceps of the reluctant diaphragm. Polypropylene sutures (zero or 1) were used to perform the plication of the diaphragm. in making a fold on itself. The plication was performed using interrupted polypropylene U-stitches; usually, it started from posterior part to the anterior part of the diaphragm. We merged every two rows with continuous polypropylene sutures. The diaphragm became tough and firm and returned to its normal position. An intercostal tube was inserted, and the thoracotomy was closed in layers.

SUMMARY:
Objectives: We aim to clarify the role of diaphragm ultrasonography (DUS) in evaluating the outcome of surgical diaphragmatic plication (SDP) in adults with symptomatic unilateral diaphragmatic paralysis (UDP).

ELIGIBILITY:
Inclusion Criteria:

- Symptomatic unilateral diaphragmatic paralysis.

Exclusion Criteria:

* Children
* Morbid obesity
* Certain neuromuscular disorders
* Previous thoracic surgical intervention on the affected
* Recurrent eventration

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: symptomatic unilateral diaphragmatic paralysis patients who underwent surgical diaphragmatic plication presented during a period from January 2015 to January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Radiological examination for diagnosis of diaphragmatic paralysis and the changes post surgical diaphragmatic plication for the management of unilateral diaphragmatic paralysis. | Chest sonography was done before operation; and follow up at one week and 6 months, through study completion, an average of 1 year .
  The radiological investigation included; chest sonography.
Respiratory functions test for evaluation of the changes post surgical diaphragmatic plication for the management of unilateral diaphragmatic paralysis. | Spirometry was done before operation; and follow up at one week and 6 months postoperatively, through study completion, an average of 1 year .
  Spirometry was done (FEV1 in %, FVC in %, FEV1/FVC in %).
Radiological examination for diagnosis of diaphragmatic paralysis and the changes post surgical diaphragmatic plication for the management of unilateral diaphragmatic paralysis. | Chest X-ray was done before operation; and follow up at one week and 6 months postoperatively, through study completion, an average of 1 year.
  The radiological investigation included; chest X-ray.

SECONDARY OUTCOMES:
Evaluation of the efficacy of surgical diaphragmatic plication and its effect on improving patients' symptoms. | the data were collected preoperatively as a baseline; one week and 6 months postoperatively.
  the clinical dyspnoea evaluation according to MRC score.

IPD SHARING:
Plan to Share IPD: No